CLINICAL TRIAL: NCT04075799
Title: A HIIT to Improve Metabolic Health in Obese Adults With Insulin Resistance
Brief Title: High-intensity Interval Training for Obese Individuals
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 restrictions.
Sponsor: University of New Mexico (Other)
Collaborators: New Mexico Inbre (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07419
Record Dates: First submitted 2019-08-13; First posted 2019-09-03 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Obesity; Insulin Resistance
Keywords: obesity; insulin resistance; high-intensity interval training
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- training (Experimental): 8 weeks using stair climbing with a frequency of thrice a week. For the first week of the stair training exercise program subjects will meet at UNM's Teaching Education Building (Stair Case 2). The following 7 weeks subjects can perform the exercise program at a staircase most convenient to them and approved by the research team. The warm-up will consist of 2 minutes of ascending and descending the stairs at a comfortable pace. The high-intensity intermittent exercise will be comprised of 6-12 x 30-seconds bout of ascending at an all-effort. A 30- seconds walking recovery will occur between the exercise bouts. After the exercise session the subject will walk during a 2-minute cool down. Every session will last between 10 to 15 minutes. The number of bouts (6-12) will be increased progressively over the weeks.
  Interventions: Other: high-intensity interval training

INTERVENTIONS:
Other: high-intensity interval training — The HIIT protocol consists of 8 weeks using stair climbing three times per week. The warm-up will consist of 2 minutes of ascending and descending the stairs at a comfortable pace. The high-intensity intermittent exercise will comprise 6-12 x 30-seconds bouts of ascending at an all-effort. A 30- seconds walking recovery will occur between the exercise bouts. Post-exercise the subject will walk during a 2-minute cool down. Every session will last between 10 to 15 minutes. The number of bouts (6-12) will be increased progressively over the weeks. The first (week 1) and final week (week 8) of the exercise program will be monitored by a trained exercise physiologist. During supervised visits, heart rate and rating of perceived exertion (OMNI scale) will be measured at the end of each bout and after active recovery. Subjects will have the option to request further monitoring if desired.

SUMMARY:
This proposal's objective is to investigate the effects of a high-intensity intermittent stair climbing program on insulin resistance in individuals with obesity and at risk of type 2 diabetes (T2D).

Obesity (defined as body mass index ≥ 30kg/m2) is a major risk factor for T2D. The connection between obesity and T2D involves the development of insulin resistance (IR). Exercise training is an effective non-pharmacological approach to prevent and treat IR. Despite the efficacy of exercise training on ameliorating IR, most individuals do not achieve the minimum recommended levels of physical activity and cite "lack of time" and difficulty in accessing exercise facilities as barriers to exercise. Proposed as a time-efficient alternative, high-intensity interval training (HIIT), which consists of short periods of high-intensity efforts alternated with brief periods of recovery, is an efficient strategy to improve IR. However, most HIIT protocols have been studied in laboratory-based settings requiring access to specialized equipment (i.e. treadmills, cycle ergometers) and are not practical for the general population. The use of high-intensity intermittent stair climbing may be a suitable exercise strategy from an accessibility perspective. With evidence to suggest improvements in IR following HIIT in individuals with obesity or T2D, the application of a similar approach using high-intensity intermittent stair climbing to directly assess changes in IR in a population at risk of T2D populations is warranted. Completion of this study will help elucidate if an easy to implement, time-efficient and low-cost exercise training program improves insulin resistance in individuals at risk of T2D.

DETAILED DESCRIPTION:
Significance The obesity epidemic is a worldwide public health problem. Recent data indicate that over 650 million adults around the world (~13%) are considered obese. Obesity is one of the major risk factors for type 2 diabetes mellitus (T2D) and 90% of T2D cases are attributable to excess fat mass. The connection between obesity and T2D is believed to be intrinsically related to insulin resistance (IR). IR is characterized by a blunted effect of insulin on decreasing circulating blood glucose at the whole-body level and/or a lower response of certain tissues to the action of insulin. For example, skeletal muscle is responsible for ~70% of insulin-stimulated postprandial glucose uptake and plays a key role in the maintenance of whole-body insulin sensitivity and glycemic homeostasis. Additionally, IR is one of the earliest detectable defects preceding hyperglycemia, present up to 10 years before diabetes is diagnosed.

Although the cause of obesity-induced IR is complex and multifactorial, the beneficial effects of exercise training in preventing and treating IR are well established. In individuals with IR, an improvement in insulin action on skeletal muscle glucose metabolism is one of the main effects induced by exercise training. For example, previous research demonstrated that a single session of exercise reduced cellular stress, which may contribute to exercise-induced increases in insulin sensitivity. Despite the efficacy of exercise training on IR, the majority of individuals do not achieve the minimum recommended levels of physical activity: 30 minutes or more of moderate intensity physical activity at least 5 days a week, or 20 minutes of vigorous physical activity at least 3 days a week, or a combination thereof, in addition to activities of daily living. Of note, lack of time and difficulty in accessing facilities for exercise are commonly cited as barriers to physical activity.

In this context, the high-intensity interval training (HIIT), which consists of short periods of intense exercise (≥ 80% of maximal heart rate) alternated with periods of active recovery or rest, is a relatively time-efficient training strategy to improve metabolic health and has been considered more enjoyable than moderate-to-vigorous intensity continuous training. HIIT increases skeletal muscle oxidative capacity and induces physiological remodeling like the changes promoted by continuous moderate-intensity aerobic training. HIIT appears effective in improving insulin sensitivity, particularly in those at risk of, or with, T2D. A previous study using 10 x of 60-seconds of cycling intervals (∼90% of maximal heart rate) interspersed with 60-seconds of active recovery, three times per week over a period of two weeks, reduced hyperglycemia and increased skeletal muscle oxidative capacity in patients with T2D. Recently published data has shown that an 8-week HIIT program resulted in lower IR in individuals with obesity and also promoted greater expression of proteins related to oxidative metabolism in skeletal muscle. Although HIIT may be an efficient option to improve insulin sensitivity and glycemic control in individuals at risk of T2D, most HIIT studies have been conducted primarily in traditional laboratory setting and may not be practical for the general population.

Innovation The common approach to study the effects of exercise are either using treadmills or cycle ergometers. These approaches have limited translation to a "real word" scenario. Among the barriers generally reported for a regular physical activity program are lack of time, difficulty in accessing facilities for exercise, and low motivation. The goal of the proposed study is to investigate the effects of a HIIT program using a suitable exercise alternative (stair climbing) on IR in individuals with obesity and at risk of T2D. Stair climbing can be considered an activity of daily living and is easily accessible. Previous studies have shown that one short bout of stair climbing (<6 min) acutely increased postprandial glucose uptake in middle-aged men with impaired glucose tolerance and older T2D subjects. Another study showed 6 weeks of a brief high intense intermittent stair climbing program was effective improving cardiorespiratory fitness in healthy individuals but did not improve IR. More recently, a preliminary study examined the effect of 6 weeks of brief intermittent stair climbing exercise on glycemic control in people with T2D. The authors reported that the protocol (3 x 1-minute bouts of repeatedly ascending and descending a single flight of stairs) was insufficient to induce improvements in glucose control. In this context, the volume was too low (approximately 50 stairs) and there was no progression of training volume over time. Additionally, the authors counted for the time descending the stairs as part of the 1-minute bout which may have reduced even more the time spent ascending the stairs. To address these limitations, the proposed study will implement a more prolonged protocol with progressive increase in exercise volume and will only count the time spent ascending the stairs. To the best of the author's knowledge, no study has tested this approach using HIIT in individuals with obesity and a risk of T2D. Findings from this study will help to translate research-based evidence to clinical practice and contribute to prevent or treat individuals at risk of T2D with a nonpharmacological and low-cost approach. This topic is within the "Cell and Organism" New Mexico - Idea Network of Biomedical Research Excellence (NM-INBRE) focus area to advance the understanding of human health.

Approach The study is an 8-wk within-subject intervention design where participants will be tested pre and post intervention. 20 participants (10 males and 10 females) will be recruited from the local community through poster advertisement and one-to-one interaction. Before agreeing to participate in the study, the participants will given written informed consent, which will be approved by the institutional review board of the local institution. Inclusion criteria include body mass index (BMI) ≥ 30 kg/m2; homeostasis model assessment for insulin resistance (HOMA-IR) ≥ 2.71; no fear of being totally submerged underwater; freedom from orthopedic injuries, diagnoses of T2D or glucose intolerance, known acute or chronic diseases, and current use of anti-inflammatory, hypoglycemic or other drugs known to affect metabolism. Subjects that meet the initial requirements will have a fasting blood draw. Individuals with altered glucose metabolism (fasting plasma glucose >126 mg/dL) will be excluded. The researchers will ensure the inclusion of males and females from differing ethnic background. The required sample size was calculated a priori based on changes in the HOMA-IR using an alpha level of 0.05 and power of 80%. Prior to exercise training, participants undergo: a fasting blood draw for blood glucose and insulin measurements, anthropometrics and body composition analysis, and a maximal graded exercise test.

The exercise training protocol consist of 8 weeks of HIIT using stair climbing with a frequency of 3 times a week, totaling 24 training sessions. For the first week of the stair training exercise program subjects will meet at UNM's Teaching Education Building (Stair Case 2). The following 7 weeks subjects can perform the exercise program at a staircase most convenient to them and approved by the research team. The warm-up will consist of 2 minutes of ascending and descending the stairs at a comfortable pace. The high-intensity intermittent exercise will be comprised of 6-12 x 30-seconds bout of ascending at an all-effort at a moderate pace. A 30- seconds walking recovery will occur between the exercise bouts. After the exercise session the subject will walk during a 2-minute cool down. Every session will last between 10 to 15 minutes. The number of bouts (6-12) will be increased progressively over the weeks. During the first (week 1) and final week (week 8) of the exercise program subjects will be monitored by a trained exercise physiologist. During these supervised visits, heart rate and rating of perceived exertion (OMNI scale) will be measured at the end of each stair climbing bout and after active recovery. Subjects will have the option to request further monitoring if desired. Weeks 2 through 7 OMNI will be self-recorded by the subjects.

Measurements Insulin resistance - After a 10-hour fast and at least 72 hours before and after the training, venous blood samples will be collected for the measurement of blood glucose and insulin. HOMA-IR (calculated by [glucose (mmol)] x [insulin (µU/ml)] ÷ 22.5) will be determined from the fasting glucose and insulin concentrations.

Anthropometric and body composition measurements - Height and body mass will be measured using an analog scale with coupled stadiometer. BMI will be calculated using height in m and body mass in kg. Relative body fat (%BF) values will be determined through underwater weighing (UWW) at measured residual lung volume. The highest 3 UWW trials ± 100 g will be averaged and used for computation of body volume. Body volume will be corrected for residual lung volume using the dry-land oxygen dilution technique so that body density can be computed and converted into %BF formula.

Maximal Oxygen Consumption - Maximal oxygen consumption will be measured using a maximal ramp graded test protocol conducted on a treadmill. The speed will be increased every 60s at an individual rate, which will be based on the participant's exercise history questionnaire (Veterans Specific Activity Questionnaire), to induce fatigue within 8 to 12 minutes. Expired gases will be analyzed using a metabolic cart. Heart rate (HR) will be recorded continuously using a HR transmitter strap (S810i series, Polar, USA).

Calculations and Statistical Analyses Data will be presented as mean ± standard deviation. A statistical software will be used for statistical analysis. The Shapiro-Wilk test will be used to analyze the data normality. Area under the curve (AUC) for insulin and glucose will be calculated using the Trapezoidal method. For study 1, a Student t test will be used to analyze the effects of training (pre vs post). For study 2, a two-way analyses of variance (ANOVA) will be used to test the effect of the two exercise protocols (factor 1 = pre and post 8 weeks of training and factor 2 = single session vs multiple sessions). If statistically significant F values are observed, a Tukey post hoc test will be performed. The alpha level is set at P ≤ 0.05 for statistical significance.

Potential problems and strategies: Dropout and compliance are limitations in exercise training interventions. The researchers will provide training session on three different times a day (early morning, afternoon and evenings) to accommodate people with different schedules. Also, participants will be compensated for time.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years,
* body mass index (BMI) equal or superior than 30 kg/m²;
* homeostasis model assessment for insulin resistance (HOMA-IR) ≥ 2.71,
* no fear of being totally submerged underwater for 2 to 10 seconds
* comfortable having blood taken from a forearm vein.

Exclusion Criteria:

* smokers,
* currently taking any medications known to impact their metabolism or immune system,
* bleeding or blood clotting disorder,
* physical injury,
* physical limitations,
* diagnostic of T2D,
* currently under the active care of a physician for any condition that may interfere with their safety.
* cardiovascular conditions (cardiac, peripheral vascular, or cerebrovascular disease),
* diseases that prevent participation in a maximal effort test without physician clearance per the American College of Sports Medicine (ACSM) guidelines (2017).
* signs and symptoms of cardiovascular disease, at rest or during physical activity, which includes pain, discomfort in the chest, neck, jaw, arms, or other areas that may result from ischemia; shortness of breath at rest or with mild exertion; dizziness or syncope; orthopnea or paroxysmal nocturnal dyspnea; ankle edema; palpitations or tachycardia; intermittent claudication; known heart murmur; or unusual fatigue or shortness of breath with usual activities.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Change in HOMA-IR concentration | Before the 8-week intervention and 72-hours after last exercise session.
  homeostasis model assessment for insulin resistance (HOMA-IR)

SECONDARY OUTCOMES:
Change in Body Composition | After a 10-hour fast and at least 72 hours before and after the training
  underwater weighing (UWW)
Change in Maximal Oxygen Consumption | After a 10-hour fast and at least 72 hours before and after the training
  maximal ramp graded test protocol on a treadmill

CONTACTS AND LOCATIONS:
Overall Officials: Fabiano Amorim, PhD, Principal Investigator — University of New Mexico
Locations (1):
- Fabiano Trigueiro Amorim, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO WHO. Obesity and overweight 2017
- [Background] Zhang L, Feng Y, List J, Kasichayanula S, Pfister M. Dapagliflozin treatment in patients with different stages of type 2 diabetes mellitus: effects on glycaemic control and body weight. Diabetes Obes Metab. 2010 Jun;12(6):510-6. doi: 10.1111/j.1463-1326.2010.01216.x. PMID 20518806
- [Background] Hossain P, Kawar B, El Nahas M. Obesity and diabetes in the developing world--a growing challenge. N Engl J Med. 2007 Jan 18;356(3):213-5. doi: 10.1056/NEJMp068177. No abstract available. PMID 17229948
- [Background] Felber JP, Golay A. Pathways from obesity to diabetes. Int J Obes Relat Metab Disord. 2002 Sep;26 Suppl 2:S39-45. doi: 10.1038/sj.ijo.0802126. PMID 12174327
- [Background] DeFronzo RA, Jacot E, Jequier E, Maeder E, Wahren J, Felber JP. The effect of insulin on the disposal of intravenous glucose. Results from indirect calorimetry and hepatic and femoral venous catheterization. Diabetes. 1981 Dec;30(12):1000-7. doi: 10.2337/diab.30.12.1000. No abstract available. PMID 7030826
- [Background] Zierath JR, Krook A, Wallberg-Henriksson H. Insulin action and insulin resistance in human skeletal muscle. Diabetologia. 2000 Jul;43(7):821-35. doi: 10.1007/s001250051457. No abstract available. PMID 10952453
- [Background] Di Meo S, Iossa S, Venditti P. Skeletal muscle insulin resistance: role of mitochondria and other ROS sources. J Endocrinol. 2017 Apr;233(1):R15-R42. doi: 10.1530/JOE-16-0598. PMID 28232636
- [Background] Keshel TE, Coker RH. Exercise Training and Insulin Resistance: A Current Review. J Obes Weight Loss Ther. 2015 Jul;5(Suppl 5):S5-003. doi: 10.4172/2165-7904.S5-003. Epub 2015 Jul 30. PMID 26523243
- [Background] Bird SR, Hawley JA. Update on the effects of physical activity on insulin sensitivity in humans. BMJ Open Sport Exerc Med. 2017 Mar 1;2(1):e000143. doi: 10.1136/bmjsem-2016-000143. eCollection 2016. PMID 28879026
- [Background] Henriksen EJ. Invited review: Effects of acute exercise and exercise training on insulin resistance. J Appl Physiol (1985). 2002 Aug;93(2):788-96. doi: 10.1152/japplphysiol.01219.2001. PMID 12133893
- [Background] de Matos MA, Ottone Vde O, Duarte TC, Sampaio PF, Costa KB, Fonseca CA, Neves MP, Schneider SM, Moseley P, Coimbra CC, Magalhaes Fde C, Rocha-Vieira E, Amorim FT. Exercise reduces cellular stress related to skeletal muscle insulin resistance. Cell Stress Chaperones. 2014 Mar;19(2):263-70. doi: 10.1007/s12192-013-0453-8. Epub 2013 Aug 22. PMID 23975543
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Background] Sherwood NE, Jeffery RW. The behavioral determinants of exercise: implications for physical activity interventions. Annu Rev Nutr. 2000;20:21-44. doi: 10.1146/annurev.nutr.20.1.21. PMID 10940325
- [Background] Korkiakangas EE, Alahuhta MA, Laitinen JH. Barriers to regular exercise among adults at high risk or diagnosed with type 2 diabetes: a systematic review. Health Promot Int. 2009 Dec;24(4):416-27. doi: 10.1093/heapro/dap031. Epub 2009 Sep 30. PMID 19793763
- [Background] Helgerud J, Hoydal K, Wang E, Karlsen T, Berg P, Bjerkaas M, Simonsen T, Helgesen C, Hjorth N, Bach R, Hoff J. Aerobic high-intensity intervals improve VO2max more than moderate training. Med Sci Sports Exerc. 2007 Apr;39(4):665-71. doi: 10.1249/mss.0b013e3180304570. PMID 17414804
- [Background] Kong Z, Fan X, Sun S, Song L, Shi Q, Nie J. Comparison of High-Intensity Interval Training and Moderate-to-Vigorous Continuous Training for Cardiometabolic Health and Exercise Enjoyment in Obese Young Women: A Randomized Controlled Trial. PLoS One. 2016 Jul 1;11(7):e0158589. doi: 10.1371/journal.pone.0158589. eCollection 2016. PMID 27368057
- [Background] Gibala MJ, Gillen JB, Percival ME. Physiological and health-related adaptations to low-volume interval training: influences of nutrition and sex. Sports Med. 2014 Nov;44 Suppl 2(Suppl 2):S127-37. doi: 10.1007/s40279-014-0259-6. PMID 25355187
- [Background] Jelleyman C, Yates T, O'Donovan G, Gray LJ, King JA, Khunti K, Davies MJ. The effects of high-intensity interval training on glucose regulation and insulin resistance: a meta-analysis. Obes Rev. 2015 Nov;16(11):942-61. doi: 10.1111/obr.12317. PMID 26481101
- [Background] Little JP, Gillen JB, Percival ME, Safdar A, Tarnopolsky MA, Punthakee Z, Jung ME, Gibala MJ. Low-volume high-intensity interval training reduces hyperglycemia and increases muscle mitochondrial capacity in patients with type 2 diabetes. J Appl Physiol (1985). 2011 Dec;111(6):1554-60. doi: 10.1152/japplphysiol.00921.2011. Epub 2011 Aug 25. PMID 21868679
- [Background] Takaishi T, Imaeda K, Tanaka T, Moritani T, Hayashi T. A short bout of stair climbing-descending exercise attenuates postprandial hyperglycemia in middle-aged males with impaired glucose tolerance. Appl Physiol Nutr Metab. 2012 Feb;37(1):193-6. doi: 10.1139/h11-140. Epub 2011 Dec 23. PMID 22196221
- [Background] Honda H, Igaki M, Hatanaka Y, Komatsu M, Tanaka S, Miki T, Suzuki T, Takaishi T, Hayashi T. Stair climbing/descending exercise for a short time decreases blood glucose levels after a meal in people with type 2 diabetes. BMJ Open Diabetes Res Care. 2016 Jul 25;4(1):e000232. doi: 10.1136/bmjdrc-2016-000232. eCollection 2016. PMID 27547414
- [Background] Allison MK, Baglole JH, Martin BJ, Macinnis MJ, Gurd BJ, Gibala MJ. Brief Intense Stair Climbing Improves Cardiorespiratory Fitness. Med Sci Sports Exerc. 2017 Feb;49(2):298-307. doi: 10.1249/MSS.0000000000001188. PMID 28009784
- [Background] Godkin FE, Jenkins EM, Little JP, Nazarali Z, Percival ME, Gibala MJ. The effect of brief intermittent stair climbing on glycemic control in people with type 2 diabetes: a pilot study. Appl Physiol Nutr Metab. 2018 Sep;43(9):969-972. doi: 10.1139/apnm-2018-0135. Epub 2018 May 2. PMID 29717900
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Wilmore JH. A simplified method for determination of residual lung volumes. J Appl Physiol. 1969 Jul;27(1):96-100. doi: 10.1152/jappl.1969.27.1.96. No abstract available. PMID 5786976
- [Background] BROZEK J, GRANDE F, ANDERSON JT, KEYS A. DENSITOMETRIC ANALYSIS OF BODY COMPOSITION: REVISION OF SOME QUANTITATIVE ASSUMPTIONS. Ann N Y Acad Sci. 1963 Sep 26;110:113-40. doi: 10.1111/j.1749-6632.1963.tb17079.x. No abstract available. PMID 14062375
- [Result] Shaw JE, Sicree RA, Zimmet PZ. Global estimates of the prevalence of diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Jan;87(1):4-14. doi: 10.1016/j.diabres.2009.10.007. Epub 2009 Nov 6. PMID 19896746